CLINICAL TRIAL: NCT03515135
Title: Metacognitive Executive Function Training for Preschool Children With ADHD - A Randomized Controlled Study
Brief Title: A Randomized Controlled Study of MEFP for Preschool Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jinsong Zhang, Director of Department of Medical Psychology, Department of Developmental Behavioral and Child Healthcare, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: XH-17-003
Record Dates: First submitted 2017-11-07; First posted 2018-05-03 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: ADHD; Child, Only
Keywords: ADHD; executive function; preschool; intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in this group will receive the "Metacognitive Executive Function Training (MEFP)" program in aiming to reduce ADHD symptoms and improve the executive function.
  Interventions: Behavioral: Metacognitive Executive Function Training
- Waiting group (No Intervention): Subjects in this group will not receive the MEFP program during the study period.

INTERVENTIONS:
Behavioral: Metacognitive Executive Function Training — Training the executive funtions of preshcool ADHD children through tasks and games repeatly but with fun. Giving the parents strategies to help the prechool ADHD childred coping the symptoms and develop EF in the reallife.
  Arms: Intervention group

SUMMARY:
The goal of this study is to provide a new, early treatment approach for preschoolers with ADHD, which could facilitate the EF developing well to achieve better outcome.

DETAILED DESCRIPTION:
ADHD in preschoolers has become established as a valid psychiatric disorder with characterized core deficits of executive function (EF). The EF impairments occurred in preschool period could persist to childhood, adolescent and adulthood, causing extensive and deep damage of individual's academic and career achievement, social function, and peer relationship. Psychostimulants remain a controversial opinion for preschoolers and appear less efficacious and more common side effects. It is very important to explore the effective nonpharmacological intervention targeting the EF deficits and appropriately tailored to young children. Therefore, the investigators conduct this randomized and controlled study to find out the therapeutic efficacy of metacognitive Executive Function Training for Preschool Children with ADHD (MEFP), and follow the subjects to observe whether the therapeutic efficacy would persist. In the mean time, the investigators also observe the factors which can influence the therapeutic efficacy. The goal of this study is to provide a new, early treatment approach for preschoolers with ADHD, which could facilitate the EF developing well to achieve better outcome.

ELIGIBILITY:
Inclusion Criteria:

1. meet both the criteria of ADHD based on the interview by the DIPA and clinical diagnosis with DSM-5;
2. full-scale IQ estimated by the Wechsler Primary and Preschool Scale of Intelligence (WPPSI) above 80;
3. their parents volunteered to participate in this study.

Exclusion Criteria:

1. child with severe mental disorder or physical disease that might interfere the assessment and intervention, such as Autistic Spectrum Disorder(ASD), schizophrenia, epilepsy, traumatic brain injury, etc.;
2. receive medication intervention for their ADHD symptoms before study;
3. parents with severe mental illness, such as schizophrenia, mood disorder (period of onset), etc..

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
The executive function of preschool child of ADHD | through the intervention completion, an average of 8 weeks
  The executive function of preschool children of ADHD assessed by neuropsychological evaluation tool NEPSY

SECONDARY OUTCOMES:
The executive function in real life of preschool child of ADHD | through the intervention completion, an average of 8 weeks
  The executive function in real life of preschool children of ADHD assessed by BRIEF
The ADHD symptoms of child | through the intervention completion, an average of 8 weeks
  The ADHD symptoms of child assessed by SNAP

CONTACTS AND LOCATIONS:
Overall Officials: Lan Shuai, Ph.D, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided